CLINICAL TRIAL: NCT05768906
Title: (DIS)AGreement of Relatives Regarding Ethical End-of-life Decisions in ICU.
Acronym: (DIS)AGREE
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: (DIS)AGREE - 2022-02
Record Dates: First submitted 2023-02-14; First posted 2023-03-15 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Cessation of Treatment; End of Life
MeSH Terms: conditions — Death | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Life-sustaining therapies limitation decision situations - observation only: For each participating center, consecutive inclusion of the first 10 life-sustaining therapies limitation decision situations from the study start date over a maximum of 12 months. Data collection for these patients especialy information concerning disagreements and even real legal conflicts on life-sustaining therapies limitation decisions between relatives and physicians.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — Observation of disagreements and even real legal conflicts on life-sustaining therapies limitation decisions between relatives and physicians

SUMMARY:
In the ICU, the vast majority of patients die following a life-sustaining therapies (LST) limitation decision. Most often, the patient is not able to express himself and has not made his wishes known beforehand, for example in the form of advance directives. The "relatives" are then the only recourse to state the patient's wishes, without any guarantee that they are aware of them. In France, the final decision is made by the physician (or the medical team) who is responsible for it. In this context, disagreements and even real legal conflicts on LST limitation decisions between relatives and physicians seem to be more and more frequent. To our knowledge, few data exist on the frequency of these disagreements over LST limitation decisions.

The main objective of this study is to evaluate the frequency of disagreements between relatives and physicians over LST limitation decisions in adult intensive care.

DETAILED DESCRIPTION:
Context In the ICU, the vast majority of patients die following a life-sustaining therapies (LST) limitation decision. Most often, the patient is not able to express himself and has not made his wishes known beforehand, for example in the form of advance directives. The "relatives" are then the only recourse to state the patient's wishes, without any guarantee that they are aware of them. In France, the final decision is made by the physician (or the medical team) who is responsible for it. In this context, disagreements and even real legal conflicts on LST limitation decisions between relatives and physicians seem to be more and more frequent. To our knowledge, few data exist on the frequency of these disagreements over LST limitation decisions.

Purpose The main objective of this study is to evaluate the frequency of disagreements between relatives and physicians over LST limitation decisions in adult intensive care.

The secondary objectives are:

* To assess the level of agreement/disagreement between family members and physicians regarding LST limitation decisions
* To assess the proportion of disagreements experienced as conflictual
* To assess the impact of the disagreement on the LST limitation decision (implementation of the decision, time between the decision and its implementation, length of hospitalization...)
* To describe possible factors that contribute to disagreement and conflict
* To describe national LST limitation decision-making practices.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive inclusion of all situations in which a life-sustaining therapies limitation decision was made
* Patients hospitalized in a French intensive care unit
* Age of the patient ≥ 18 years
* If relatives are present, age of at least one of the relatives ≥ 18 years NB: situations of "non-re-admission" decisions in intensive care are not taken into account in the inclusion criteria.

Exclusion Criteria:

* Minor patient
* Patient under guardianship
* Conscious patient, able to express himself/herself and able to decide jointly with the medical team
* Patient for whom a life-sustaining therapies limitation decision was already made prior to ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Life-sustaining therapies limitation decision is made (during the study)
Sampling Method: Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Frequency of disagreements - Using linkert scale | At the latest by may 31, 2024
  Evaluate the frequency of disagreements between relatives and physicians over LST limitation decisions in adult intensive care. A linkert scale will be used to cote the disagreements and will be completed by the investigator.

SECONDARY OUTCOMES:
Level of agreement/disagreement - Using linkert scale | At the latest by may 31, 2024
  To assess the level of agreement/disagreement between family members and physicians regarding life-sustaining therapies limitation decisions. A linkert scale will be used to cote the level of agreement/disagreement and will be completed by the investigator. Data will be expressed as numbers and percentages or medians and interquartile ranges. The data will be compared by the appropriate non-parametric tests.
Proportion of disagreements experienced as conflictual - Using linkert scale | At the latest by may 31, 2024
  To assess the proportion of disagreements experienced as conflictual. A linkert scale will be used to cote the level of Proportion of disagreements experienced as conflictual and will be completed by the investigator. Data will be expressed as numbers and percentages or medians and interquartile ranges. The data will be compared by the appropriate non-parametric tests.
Impact of the disagreement on the life-sustaining therapies limitation decision. Evaluation by questionnary. | At the latest by may 31, 2024
  To assess the impact of the disagreement on the life-sustaining therapies limitation decision. Questionnary will be completed by the investigator.Data will be expressed as numbers and percentages or medians and interquartile ranges. The data will be compared by the appropriate non-parametric tests.
Factors identification | At the latest by may 31, 2024
  To describe possible factors that contribute to disagreement and conflict. Data will be expressed as numbers and percentages or medians and interquartile ranges. The data will be compared by the appropriate non-parametric tests
Description of national practices - Aggregation of responses from all sites | At the latest by may 31, 2024
  To describe national life-sustaining therapies limitation decision-making practices.
  Aggregation of responses to questions of the CRF from all sites Data will be expressed as numbers and percentages or medians and interquartile ranges. The data will be compared by the appropriate non-parametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael Giabicani, MD, Study Chair — Hôpital Beaujon - 100 boulevard du Général Leclerc - 92110 Clichy
Locations (23):
- France (23):
  - CH d'Aurillac (CH Henri Mondor), Aurillac
  - Hôpital Saint Camille, Bry-sur-Marne
  - CHU de Clermont Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Beaujon - Réanimation chirurgicale polyvalente, Clichy
  - Hôpital Beaujon - Réanimation hépato-digestive, Clichy
  - CH de Dieppe, Dieppe
  - CHU de Dijon, Dijon
  - Hôpital Simone Veil- Eaubonne, Eaubonne
  - CH de Grasse, Grasse
  - GHEF (Grand Hôpital de l'Est Francilien)-Site de Marne la Vallée, Jossigny
  - CHU de Grenoble-Alpes, La Tronche
  - CH de Lens, Lens
  - CHU de Montpellier - Gui de Chauliac, Montpellier
  - Hôpital Lariboisière_APHP - Réanimation Chirurgicale Polyvalente, Paris
  - Institut Mutualiste Montsouris -, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital privé Claude Galien, Quincy-sous-Sénart
  - CHU de Reims - Réanimation chirurgicale, Reims
  - CHU de Toulouse-Rangueil - Réanimation Polyvalente, Toulouse
  - CHBA Vannes-Auray, Vannes
  - CH Versailles, Versailles
  - HIA Robert Picqué, Villenave-d'Ornon
  - Médipôle Lyon Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: Undecided